CLINICAL TRIAL: NCT03193021
Title: AMBULATE: Multi-center, RCT for Safety & Efficacy of Cardiva Mid-Bore Venous VCS v. Manual Compression to Close Femoral Venotomies After Catheter-based Interventions Via 6-12F ID Sheaths With Single or Multiple Access Sites Per Limb
Brief Title: AMBULATE: Cardiva Mid-Bore VVCS vs. Manual Compression for Multiple Femoral Venous Access Sites, 6 - 12F ID
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cardiva Medical, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PTL 0508
Record Dates: First submitted 2017-06-16; First posted 2017-06-20 (Actual); Results first posted 2020-02-05 (Actual); Last update posted 2023-03-10 (Actual); Status verified 2023-02

CONDITIONS: Surgical Wound
Keywords: vessel closure; venous access site; femoral venotomy; medium bore; multiple access sites
MeSH Terms: conditions — Surgical Wound

STUDY DESIGN:
Intervention Model Description: Subjects randomized in 1:1 fashion to either Cardiva Mid-Bore Venous Vascular Closure Device (VVCD) or manual compression for multiple venous access site hemostasis
Who Masked: Outcomes Assessor
Masking Description: Data Safety Monitoring Committee will adjudicate endpoint events, blinded to treatment assignment when possible
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- Cardiva Mid-Bore VVCS (Experimental): Cardiva Mid-Bore VVCS will be used to close all femoral venous access sites at the end of the case.
  Interventions: Device: Cardiva Mid-Bore VVCS
- Manual Compression (Active Comparator): Direct manual compression to the access sites will be used to close all femoral venous access sites at the end of the case.
  Interventions: Other: Manual compression

INTERVENTIONS:
Device: Cardiva Mid-Bore VVCS — The device will be used to close all femoral venous access sites at the end of the case, which range from 3 - 4 access sites per patient.
  Arms: Cardiva Mid-Bore VVCS
Other: Manual compression — Manual compression will be used to achieve hemostasis in all femoral venous access sites when the sheaths are pulled, which range from 3-4 access sites per patient.
  Arms: Manual Compression

SUMMARY:
The objective of the trial is to demonstrate the safety and effectiveness of the Cardiva Mid-Bore Venous Vascular Closure System (VVCS) in sealing femoral venous access sites and providing reduced times to ambulation (TTA) compared with manual compression at the completion of catheter-based procedures performed through 6 - 12 Fr introducer sheaths.

DETAILED DESCRIPTION:
A prospective, randomized, controlled multi-center clinical trial designed to evaluate the safety and effectiveness of the study device in sealing multiple femoral venous access sites and providing reduced times to ambulation compared with manual compression at the completion of catheter-based procedures performed through 6 - 12 Fr introducer sheaths.

Only patients with multiple access sites will be enrolled in order to support the desired indication. Randomization will be stratified to account for patients with varying numbers of access sites in a 1:1 treatment device to control arm ratio to ensure treatment and control arms have the same proportion of access sites/patient, i.e. 3 access sites/patient vs. 4 access sites/patient.

ELIGIBILITY:
Inclusion Criteria:

* Acceptable candidate for an elective, non-emergent catheter-based procedure via the common femoral vein(s) using a 6 to 12 Fr inner diameter introducer sheath, with a minimum of 3 and maximum of 4 femoral venous access sites, and a maximum of 2 access sites/leg
* Anticipated prolonged bedrest (5 hours or more) and / or overnight stay

Exclusion Criteria:

* Active systemic or cutaneous infection, or inflammation in vicinity of the groin
* Pre-existing immunodeficiency disorder or chronic use of high dose systemic steroids
* Know history of bleeding diathesis, coagulopathy, hypercoagulability or platelet count < 100,000 cells/mm3
* Severe co-existing morbidities with life expectancy less than 12 months
* Femoral arteriotomy or femoral venotomy in < 10 days, or with any known vascular complications or residual hematoma, or with use of an intravascular closure device w/in previous 30 days
* Planned femoral venous or arterial access within next 30 days
* History of DVT, pulmonary embolism or thrombophlebitis
* Significant anemia or renal insufficiency
* BMI > 45 kg/m2 or < 20 kg/m2
* Unable to routinely walk at least 20 ft. without assistance
* LMWH within 8 hours before or after procedure
* Access site-specific eligibility criteria to exclude problems with gaining access or location of sheath; < 6 Fr or > 12 Fr inner diameter sheath use; obvious bleeding complications or tissue tract estimated to be < 2.5 cm deep

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 204 (Actual)
Dates: Start 2017-09-20 (Actual); Primary Completion 2018-04-13 (Actual); Study Completion 2018-04-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Natale, MD, Principal Investigator — Texas Cardiac Arrhythmia Research Foundation; Steve Compton, MD, Principal Investigator — Alaska Heart Institute; Mintu Turakhia, MD, Study Director — Stanford Center for Clinical Research
Locations (13):
- United States (13):
  - Alaska Heart & Vascular, Anchorage, Alaska
  - Mercy General Hospital, Sacramento, California
  - Stanford University Hospital, Stanford, California
  - Medstar Washington Hospital Center, Washington D.C., District of Columbia
  - Emory St. Joseph's Hospital, Atlanta, Georgia
  - University of Chicago, Chicago, Illinois
  - Advocate Christ Medical Center, Oak Lawn, Illinois
  - The Valley Hospital, Ridgewood, New Jersey
  - Mount Sinai Hospital, New York, New York
  - Centennial Medical Center, Nashville, Tennessee
  - Texas Cardiac Arrhythmia Research Foundation, Austin, Texas
  - Intermountain Health Care, Murray, Utah
  - University of Utah Health Sciences Center, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Natale A, Mohanty S, Liu PY, Mittal S, Al-Ahmad A, De Lurgio DB, Horton R, Spear W, Bailey S, Bunch J, Musat D, O'Neill P, Compton S, Turakhia MP; AMBULATE Trial Investigators. Venous Vascular Closure System Versus Manual Compression Following Multiple Access Electrophysiology Procedures: The AMBULATE Trial. JACC Clin Electrophysiol. 2020 Jan;6(1):111-124. doi: 10.1016/j.jacep.2019.08.013. Epub 2019 Oct 30. PMID 31971899

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Cardiva Mid-Bore VVCS | Manual Compression
Started | 100 | 104
Completed | 99 | 103
Not Completed | 1 | 1
Not completed — Lost to Follow-up | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cardiva Mid-Bore VVCS | Manual Compression | Total
Number analyzed (Participants) | 100 | 104 | 204
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.5 (11.6) | 63.4 (11.1) | 62.5 (11.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 33 | 40 | 73
  Male | 67 | 64 | 131
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 6 | 9
  Not Hispanic or Latino | 97 | 95 | 192
  Unknown or Not Reported | 0 | 3 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 3 | 0 | 3
  Asian | 2 | 1 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 6 | 4 | 10
  White | 86 | 93 | 179
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 3 | 6 | 9
Region of Enrollment [Number; unit: participants]
  United States | 100 | 104 | 204
BMI [Mean (Standard Deviation); unit: kg/m^2] | 29.5 (4.5) | 29.7 (5.2) | 29.6 (4.9)

OUTCOME MEASURES:

1. Primary Outcome: Time to Ambulation (TTA)
Description: Elapsed time between removal of the final Mid-Bore VVCS device (treatment arm) or removal of final sheath (control arm) and when subject stands and walks 20 feet without evidence of venous re-bleeding from the femoral access site.
Time Frame: Post-procedure, usually within 6 hours
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Cardiva Mid-Bore VVCS | Manual Compression
Number analyzed (Participants) | 100 | 104
hours | 2.8 (1.3) | 6.1 (1.6)

2. Primary Outcome: Major Venous Access Site Closure-related Complications, Number of Limbs With Each Event
Description: Rate of combined major venous access site closure-related complications. The method used to determine what would be considered "major" venous access site closure-related complications are those complications which were attributed directly to the closure method used for the access site at the end of the procedure.
Time Frame: 30 +/- 7 days post-procedure
Population: Major Venous Access Site Closure-Related Complications, Number of Limbs with Each Event
Measure: Number (95% Confidence Interval); unit: major complications
Units Other Than Participants: Number of Limbs
Arm/Group | Cardiva Mid-Bore VVCS | Manual Compression
Number analyzed (Participants) | 100 | 104
Number analyzed (Number of Limbs) | 199 | 209
major complications | 0 [-0.02 to 0.04] | 0 [-0.02 to 0.04]

3. Secondary Outcome: Minor Venous Access Site Closure-related Complications, Number of Limbs With Each Event
Description: Rate of combined minor venous access site closure-related complications. The method used to determine what would be considered "minor" venous access site closure-related complications are those complications which were attributed directly to the closure method used for the access site at the end of the procedure.
Time Frame: 30 +/- 7 days post-procedure
Population: Combined Venous Access Site Closure-Related Complications, As Reported, Number of Limbs with Each Event
Measure: Number; unit: minor complications
Units Other Than Participants: Number of Limbs
Arm/Group | Cardiva Mid-Bore VVCS | Manual Compression
Number analyzed (Participants) | 100 | 104
Number analyzed (Number of Limbs) | 199 | 209
minor complications | 2 | 5

4. Secondary Outcome: Time to Discharge Eligibility (TTDE)
Description: Elapsed time between removal of the final Mid-Bore VVCS device (treatment arm) or removal of final sheath (control arm) and when subject is eligible for discharge based solely on assessment of the access site
Time Frame: Prior to hospital discharge, usually within 24 hours
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Cardiva Mid-Bore VVCS | Manual Compression
Number analyzed (Participants) | 100 | 104
hours | 3.1 (1.3) | 6.5 (1.9)

5. Secondary Outcome: Time to Hemostasis (TTH)
Description: Elapsed time between removal of the final Mid-Bore VVCS device (treatment arm) or removal of final sheath (control arm) and first observed and confirmed venous hemostasis, for each access site.
Time Frame: Post-procedure, usually within 3 hours
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Cardiva Mid-Bore VVCS | Manual Compression
Number analyzed (Participants) | 100 | 104
minutes | 6.1 (3.7) | 13.7 (6.5)

6. Secondary Outcome: Time to Discharge (TTD)
Description: Elapsed time between removal of the final Mid-Bore VVCS device (treatment arm) or removal of final sheath (control arm) and when subject is discharged
Time Frame: Prior to hospital discharge, usually within 24 hours
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Cardiva Mid-Bore VVCS | Manual Compression
Number analyzed (Participants) | 100 | 104
hours | 21.8 (13.4) | 21.8 (9.5)

7. Secondary Outcome: Time to Closure Eligibility (TTCE)
Description: Elapsed time between removal of the last procedural device for the index procedure and removal of the first Mid-Bore VVCS device (treatment arm) or removal of first sheath (control arm)
Time Frame: Post-procedure, usually within 6 hours
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Cardiva Mid-Bore VVCS | Manual Compression
Number analyzed (Participants) | 100 | 104
minutes | 10.5 (6.0) | 37.6 (33.2)

8. Secondary Outcome: Total Post-Procedure Time (TPPT)
Description: Elapsed time between removal of the last procedural device for the index procedure and when the subject is able to successfully ambulate
Time Frame: Post-procedure, usually within 6 hours
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Cardiva Mid-Bore VVCS | Manual Compression
Number analyzed (Participants) | 100 | 104
hours | 3.1 (1.3) | 6.8 (1.7)

9. Secondary Outcome: Number of Participants With Procedure Success
Description: Attainment of final hemostasis at all venous access sites and freedom from major venous access site closure-related complications
Time Frame: 30 +/- 7 days post-procedure
Measure: Count of Participants; unit: Participants
Arm/Group | Cardiva Mid-Bore VVCS | Manual Compression
Number analyzed (Participants) | 100 | 104
Participants
  Study Subjects | 98 | 103
  LTF | 2 | 1

10. Secondary Outcome: Number of Access Sites With Device Success
Description: Ability to deploy the delivery system, deliver the collagen, and achieve hemostasis with the Mid-Bore VVCS (per access site analysis, treatment arm only)
Time Frame: Procedural, usually within 15 minutes of enrollment
Population: Number of access sites where device insertion was attempted.
Measure: Number; unit: Successful Femoral Access Sites
Units Other Than Participants: Femoral Access Sites
Arm/Group | Cardiva Mid-Bore VVCS
Number analyzed (Participants) | 100
Number analyzed (Femoral Access Sites) | 363
Successful Femoral Access Sites | 351

ADVERSE EVENTS:
Time Frame: 30 days (± 7 days)
Arm/Group | Cardiva Mid-Bore VVCS | Manual Compression
All-Cause Mortality (participants affected / at risk) | 0/100 | 0/104
Serious Adverse Events (participants affected / at risk) | 9/100 | 2/104
Other Adverse Events (participants affected / at risk) | 0/100 | 0/104
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cardiva Mid-Bore VVCS (N=100) | Manual Compression (N=104)
POST ABLATION -SVT/ AFLUTTER (Cardiac disorders) | 1 (1) | 0 (0)
ACUTE KIDNEY INSUFFICIENCY (Renal and urinary disorders) | 1 (1) | 0 (0)
ACUTE DIASTOLIC HEART FAILURE EXACERBATION (Cardiac disorders) | 1 (1) | 0 (0)
Arterial Perforation - non-access site-related (Cardiac disorders) | 1 (1) | 0 (0)
CHEST PAIN (Cardiac disorders) | 1 (1) | 0 (0)
CHF EXACERBATION (Cardiac disorders) | 0 (0) | 1 (1)
FLUID OVERLOAD (Surgical and medical procedures) | 1 (1) | 0 (0)
HYPOTENSION (Cardiac disorders) | 1 (1) | 0 (0)
NEW ONSET A-FLUTTER (Cardiac disorders) | 1 (1) | 0 (0)
PERICARDIAL EFFUSION (Cardiac disorders) | 1 (1) | 0 (0)
PERICARDITIS (Cardiac disorders) | 0 (0) | 1 (1)
PNEUMONIA (Infections and infestations) | 1 (1) | 0 (0)
POST ABLATION FEVER (Surgical and medical procedures) | 1 (1) | 0 (0) — Procedural Complication
Pseudoaneurysm requiring thrombin/fibrin adhesive injection or ultrasound-guided compression (Surgical and medical procedures) | 1 (1) | 0 (0)
Access site hematoma < 6 cm (Surgical and medical procedures) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2017-12-22): https://cdn.clinicaltrials.gov/large-docs/21/NCT03193021/Prot_SAP_ICF_000.pdf